CLINICAL TRIAL: NCT04948645
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Assess Safety, Tolerability, and Pharmacokinetics Following Multiple Doses of Fosigotifator in Subjects With Amyotrophic Lateral Sclerosis Followed by an Active Treatment Extension
Brief Title: A Phase 1 Study to Investigate the Safety and Pharmacokinetics of Fosigotifator in Patients With Amyotrophic Lateral Sclerosis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Company Decision
Sponsor: AbbVie (Industry)
Collaborators: Calico Life Sciences LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M20-405
Record Dates: First submitted 2021-06-23; First posted 2021-07-02 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: ALS; Amyotrophic Lateral Sclerosis
Keywords: Fosigotifator; ABBV-CLS-7262
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Fosigotifator Low Dose (Active Comparator)
  Interventions: Drug: Fosigotifator
- Fosigotifator Medium Dose (Active Comparator)
  Interventions: Drug: Fosigotifator
- Fosigotifator High Dose (Active Comparator)
  Interventions: Drug: Fosigotifator
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fosigotifator — Oral
  Other Names: ABBV-CLS-7262
  Arms: Fosigotifator High Dose; Fosigotifator Low Dose; Fosigotifator Medium Dose
Drug: Placebo — Oral
  Arms: Placebo

SUMMARY:
Fosigotifator is an investigational drug being researched for the treatment of Amyotrophic Lateral Sclerosis. This is an up to 156-week, 2-part study. Part 1 will be a 4-week, randomized, double-blind, placebo-controlled study; Part 2 will be up to a 152-week active treatment extension (ATE) during which all subjects will receive Fosigotifator.

ELIGIBILITY:
Inclusion Criteria:

* Must have an identified, reliable caregiver.
* Confirmed diagnosis of Familial Amyotrophic Lateral Sclerosis (ALS) or Sporadic ALS.
* First ALS symptoms occurred <= 36 months before screening.
* Able to swallow solids.
* No known active COVID-19 infection at screening.
* Slow vital capacity (SVC) >= 50% predicted value (for sex, age, ethnic origin, and height) at screening.
* If taking concomitant standard-of-care medications approved for the treatment of ALS (or their components), subjects must be on a stable dose of the medication(s) for >30 days prior to Baseline in order to enter the study. For edaravone, a stable dose is defined by having completed 2 treatment cycles prior to Baseline.

Exclusion Criteria:

* History of dementia/severe cognitive problems at screening.
* History of clinically significant medical conditions (other than ALS) or any other reason, including any physical, psychological, or psychiatric condition that, in the opinion of the Investigator, would compromise the safety or interfere with the subject's participation in the study, or would make the subject an unsuitable candidate to receive study drug, or would put the subject at risk by participating in the study.
* History of abnormal screening laboratory or imaging results that, in the opinion of the Investigator, are indicative of any significant cardiac, endocrinologic, hematologic, hepatic, immunologic, infectious, metabolic, urologic, pulmonary, gastrointestinal, dermatologic, psychiatric, renal, neurologic, and/or other major disease that would preclude administration of Fosigotifator.
* Documented active or suspected malignancy or history of any malignancy within the last 5 years except for successfully treated non-melanoma skin cancer or localized carcinoma in situ of the cervix.
* If female, is known to be pregnant, breastfeeding, considering becoming pregnant, or donating/banking eggs during the study or within 30 days or >5 half-lives (whichever is longer) after the last dose of study drug.
* If male, plans to donate sperm or father a child during the study or within 30 days after the last dose of study drug.
* Known to have received any investigational product within 30 days or 5 half-lives of the drug (whichever is longer) prior to the first dose of study drug or is currently enrolled in another clinical study.
* History of Fosigotifator use prior to participation in this study.
* Recent (within 6 months prior to Screening) history of drug or alcohol abuse.
* Previous participation in a stem cell clinical study for treatment of ALS.
* Current or anticipated use of diaphragmatic pacing during the study period.
* Tracheostomy or use of non-invasive ventilatory support >= 22 hours a day.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2021-09-22 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability | Baseline Up to Approximately Day 28
  Number of patients with treatment-related adverse events as assessed by CTCAE v4.03
Pharmacokinetics | Baseline Up to Approximately Day 28
  Maximum Plasma Concentration [Cmax]
Pharmacokinetics | Baseline Up to Approximately Day 28
  Area Under the Curve [AUC]

SECONDARY OUTCOMES:
CSF Pharmacokinetics | Baseline Up to Approximately Day 28
  Concentration at steady state in CSF
Safety and Tolerability | Baseline Up to Approximately Week 156
  Number of patients with treatment-related adverse events as assessed by CTCAE v4.03

CONTACTS AND LOCATIONS:
Locations (14):
- United States (7):
  - UC Irvine Health ALS and Neuromuscular Center, Irvine, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Forbes Norris MDA/ALS Research and Treatment Center, San Francisco, California
  - Mayo Clinic, Jacksonville, Florida
  - Johns Hopkins ALS Clinical Trials Unit, Baltimore, Maryland
  - Healey & AMG Center for ALS Research, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
- Canada (7):
  - University of Calgary - Heritage Medical Research Clinic, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - Stan Cassidy Centre for Rehabilitation, Fredericton, New Brunswick
  - London Health Sciences Centre, London, Ontario
  - Sunnybrook Research Institute, Toronto, Ontario
  - Centre Hospitalier de l'Universite de Montreal (CHUM), Montreal, Quebec
  - Montreal Neurological Institute and Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No